CLINICAL TRIAL: NCT00140075
Title: Phase III, Randomized Study Of Epirubicin/Cyclophosphamide Followed By Taxane (Sequential Chemotherapy) Versus Epirubicin/Taxane (Concurrent Chemotherapy) As Adjuvant Treatment For Operable, Node-Positive Breast Cancer
Brief Title: Adjuvant Epirubicin/Cytoxan Followed By A Taxane VS. Epirubicin/Taxane As Treatment For Node-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 378-ONC-0030-184
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): ET (8 cycles)
  T = docetaxel or paclitaxel
  Interventions: Drug: Epirubicin with a Taxane
- A (Experimental): EC (4 cycles) followed by T (4 cycles) for a total of 8 cycles
  T = docetaxel or paclitaxel
  Interventions: Drug: Epirubicin with Cyclophosphamide, followed by a Taxane

INTERVENTIONS:
Drug: Epirubicin with Cyclophosphamide, followed by a Taxane — Epirubicin = 90 mg/m2 Cyclophosphamide = 600 mg/m2
  Followed by a taxane; paclitaxel = 175 mg/m2 or docetaxel = 75 mg/m2
  Other Names: Epirubicin, ellence,
  Arms: A
Drug: Epirubicin with a Taxane — Epirubicin = 75 mg/m2 per cycle
  Taxane = paclitaxel = 175 mg/m2 or docetaxel = 75 mg/m2
  Other Names: Epirubicin, ellence,
  Arms: B

SUMMARY:
The purpose of this study is to compare two combinations of drugs, epirubicin given with a taxane (ET) or epirubicin given with cyclophosphamide (cytoxan) and followed by a taxane to see if one of the combinations is better at preventing or delaying the time for breast cancer recurrence and death after 3 years. The study will also evaluate the side effects of both treatment combinations.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer Stage T1-3, N1, M0
* Suitable candidate for anthracycline-containing adjuvant chemotherapy

Exclusion Criteria:

* Evidence of residual tumor following surgery, or metastatic disease
* Received prior therapy for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2000-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Disease free survival at 3 years | 3 years

SECONDARY OUTCOMES:
Assess safety in both treatment arms at 3 years | 3 years
Compare overall survival between the 2 treatment arms at 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (52):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Fountian Valley, California
  - Pfizer Investigational Site, Gilroy, California
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Soquel, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Lecanto, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Shores, Florida
  - Pfizer Investigational Site, Port Saint Lucie, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Belleville, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Harper Woods, Michigan
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Mount Holly, New Jersey
  - Pfizer Investigational Site, Willingboro, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Lawton, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Lemoyne, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Portsmouth, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=378-ONC-0030-184&StudyName=Adjuvant%20Epirubicin/Cytoxan%20Followed%20By%20A%20Taxane%20VS.%20Epirubicin/Taxane%20As%20Treatment%20For%20Node-Positive%20Breast%20Cancer